CLINICAL TRIAL: NCT01456182
Title: Phase 1B- Open Label Dose-Ranging Study of Oral AFX-2 in Adults With Chronic Lymphocytic Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Afexa Life Sciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: AFX-2-2010-1
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dose arm 1 (Other)
  Interventions: Drug: AFX-2
- Dose arm 2 (Other)
  Interventions: Drug: AFX-2
- Dose arm 3 (Other)
  Interventions: Drug: AFX-2
- Dose arm 4 (Other)
  Interventions: Drug: AFX-2
- Dose arm 5 (Other)
  Interventions: Drug: AFX-2

INTERVENTIONS:
Drug: AFX-2 — Dose level 1
  Arms: Dose arm 1
Drug: AFX-2 — Dose level 2
  Arms: Dose arm 2
Drug: AFX-2 — Dose level 3
  Arms: Dose arm 3
Drug: AFX-2 — Dose level 4
  Arms: Dose arm 4
Drug: AFX-2 — Dose level 5
  Arms: Dose arm 5

SUMMARY:
This trial will assess the tolerability and safety of AFX-2 over a range of five dose levels in adults with low-, intermediate- or high-risk Chronic Lymphocytic Leukemia (CLL). The trial will also determine the impact of dose on quality of life indices and on biological and immune responses, and will assess if there is a maximum tolerated dose and/or dose-limiting toxicity in this study population.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women >18 years of age
2. Diagnosis of CLL per NCI Working Group Criteria; with phenotypic evidence (i.e.. flow cytometry or bone marrow biopsy) of chronic lymphocytic leukemia (MEDDRA Code - 10008960; ICD-O3-9823)
3. Disease meets criteria for low-risk (Rai Stage 0), intermediate-risk (Rai Stage I- II), or high-risk (Rai Stage III-IV) disease
4. Life expectancy of ≥ 3 months at Screening.
5. ECOG performance status 0-3
6. Laboratory parameters (taken < 14 days of Study Day 0):

   * Hematologic parameters: Hemoglobin > 9 gm/dL (stable, not dropping); Absolute Granulocyte Count (AGC) > 1.0 x 109/L; Platelets > 50 x 109/L; not requiring immediate transfusion.
   * Coagulation: PT/PTT/INR: ± 10% of NL for lab; INR: 1.0-1.43
   * BUN < 40; serum Creatinine ≤ 2.0 mg/dL, OR Creatinine Clearance > 90 mL/min/1.73m2 IF serum Creatinine > 2.0 mg/dL
   * Liver function tests (AST, ALT, ALP, LDH): < 2.5 x institutional ULN; Total bilirubin: < 2.0 x institutional ULN
   * Human Immunodeficiency Virus (HIV) negative
   * Pregnancy test: negative urine pregnancy test for females of child-bearing potential,
7. Free of disease from prior malignancy/ies for > 2 years, except for basal cell or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix or breast.
8. If not surgically sterile, or post-menopausal (> 12 months with no menstrual flow), willing to practice birth control (barrier + contraception) throughout duration of study.
9. Able and willing to swallow capsules.
10. Willing to limit alcohol intake during the study treatment period.
11. Willing to sign the informed consent.

Exclusion Criteria:

1. Lymphoproliferative disease other than CLL
2. Prior use of the test article (AFX-2), or ginseng-containing products (American, Asian, etc.) ≤ 1 year prior to study entry.
3. Known allergy to the test article or ginseng-containing products
4. Active infection requiring systemic treatment
5. Prior or current therapy:

   * Splenectomy.
   * Currently requiring anticoagulant therapy
   * Requiring active treatment for B-CLL or ≤ 28 days post-treatment for B-CLL or other condition requiring: chemotherapy, radiation therapy, monoclonal antibodies, systemic steroids, antihistamines or non-steroidal anti-inflammatory drugs, including ibuprofen, indomethacin, COX-2 inhibitors etc.
   * ≤ 10 days: non-steroidal hormonal therapy (other than for contraception or thyroid)
   * ≤ 10 days: antibiotic prophylaxis
   * History of therapy with immunological reagents, such as allogeneic bone marrow transplant, monoclonal antibody therapy, intravenous immunoglobulin, or hematopoietic stem cell transplantation. (Note: Immunotherapy for allergies is permitted as long as the last treatment was both (a) prior to the CLL diagnosis and (b) > 5 years prior to trial enrollment.)
   * < 90 days post treatment with chlorambucil
   * < 90 days post general anesthesia
6. Uncontrolled intercurrent condition, including, but not limited to, cardiovascular, pulmonary, renal, hepatic, GI, GU, neurologic, metabolic, psychiatric, etc.
7. Current or prior investigational product or procedure < 56 days preceding study entry (Baseline -Visit 2; Study Day 0).
8. Unwilling to discontinue use of nonprescription (OTC), nutritional or dietary supplements during the study period (as further defined by protocol).
9. Pregnant, lactating.
10. Any condition, personal or social situation that precludes or limits the ability of the participant to provide informed consent or comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability will be assessed based on the incidence, duration and intensity of adverse events | 0-8 weeks
  Adverse events will be graded according to NCI-CTC v4.
Safety and tolerability will also be determined by assessing any changes in study test results from baseline values | 1 week, 4 weeks, 8 weeks
  Study tests that will determine safety include vital signs, clinical laboratory tests (hematology, serum chemistries, coagulation, urinalysis) and 12-lead EKG

SECONDARY OUTCOMES:
Quality of life indices | 1 week, 4 weeks, 8 weeks
Maximum tolerated dose and/or dose-limiting toxicity | 1 week, 4 weeks, 8 weeks
Biological and immune responses | 1 week, 4 weeks, 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Leslie R Ellis, MD, Principal Investigator — Wake Forest University Health Sciences Center
Locations (3):
- United States (3):
  - Saint Jospeh Mercy Health System, Ann Arbor, Michigan
  - Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina
  - Cancer Center of the Carolinas, Greenville, South Carolina